CLINICAL TRIAL: NCT05794347
Title: Effects of Vertical Sitting Versus Supine Lying Traction on Pain, Range of Motion and Function in Patients With Chronic Radicular Low Back Pain
Brief Title: Traction in Vertical Sitting Position Versus Supine Lying Position in Patients of Chronic Radicular Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0116
Record Dates: First submitted 2023-03-15; First posted 2023-04-03 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
Keywords: low back pain; Chronic pain; Traction
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Traction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Vertical sitting traction) (Experimental): This session will be followed by the application of the continuous mechanical traction in the vertical sitting position with a belt around the chest. A total of 30 minutes session per day with 5 sessions per week for 12 weeks will be provided to the participants in this group
  Interventions: Other: Traction
- Group-B (supine lying traction) (Active Comparator): Following the conventional treatment, continuous mechanical traction will be applied in the supine lying position with a traction force equal to 50% of the total body weight. A total of 20 minutes session per day with 5 sessions per week will be provided to the participants in group B.
  Interventions: Other: Traction

INTERVENTIONS:
Other: Traction — Continuous mechanical traction will be applied to the lumbar area in 2 different positions.

SUMMARY:
The primary objective of the study is to determine the effects of vertical sitting versus supine lying traction on pain, range of motion, and function in patients with chronic radicular low back pain (CRLBP). CRLBP is one of the major types of lower back pain and causes significant disability and reduction in quality of life in the human population. The study will be a randomized controlled trial and the study setting will be Al-Barkat Hospital Gojra . A total of 30 participants will be selected randomly employing a non-probability convenient sampling technique. Two experimental groups will be made. Group A will be given vertical traction in a sitting position and Group B will be given traction in supine lying. Both groups will receive baseline physiotherapy treatment which includes Hot-pack, TENS, and ultrasound. The Numeric Pain Rating Scale (NPRS) and Oswestry Disability Index (ODI) will be used as outcome-measuring tools for pain intensity and functional disability respectively. An inclinometer will be used to measure ROM. Measures will be taken at (0, 4th, 8th, and 12th week). Data will be analyzed by using parametric/non-parametric tests after assessing the normality. SPSS version 28.

DETAILED DESCRIPTION:
CRLBP of the lumbosacral region is a disorder that is closely linked with socioeconomic consequences. The incidence of lower back pain among workers is approximately 13%. Out of which, CRLBP is responsible for 11%. In the lumbosacral region, radicular pain has an occurrence rate of 10 % to 25%. Key interventions by physical therapists involve pain relieving modalities, stretching, muscle conditioning, lumbar traction, and awareness about correct postures that lead to useful exercises. As the reason behind the radicular low back pain is the spinal nerve compression due to the spinal canal impingement, the lumbar traction lightens the pain through vertebral separation producing decompression on the pressed nerve. Radicular low back pain shows diverse symptoms, it can be self-limiting, staying only for a short interval with no aftereffects, or can be a key concern behind long-term disability and work loss.

The narrative on the effectiveness of vertical traction as a component of physical therapy modalities is contradictory. Despite the fact that lumbar traction has been preferred over other methods for the treatment of lumbar disk disorders, it is usually not advised in the treatment of acute low back pain because of the efficiency of more active treatment options.

The aim of the study is to determine the effects of vertical sitting versus supine lying traction on pain, range of motion, and function in patients with radicular low back pain. This study may help physiotherapists to have an estimate of the best possible position for applying traction in patients with radicular low back pain. The conclusion of this study might provide therapists with an optimum traction treatment protocol for CRLBP.

ELIGIBILITY:
Inclusion Criteria:

* Both genders have an age range between 20-50 years.

  * Chronicity of radicular low back pain for at least 3 months
  * Capable of attending physiotherapy sessions regularly (5 times a week for 12 weeks)

Exclusion Criteria:

* Patients with indications of spinal cord involvement (For instance; Urine or Fecal incontinency, Lack of sensation, or Limb paralysis
* Pregnant females will not be included.
* Patients with a background of spinal trauma
* Patients presenting a history of systemic disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | follow up at 12th week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. It has 10 different sections. For each section the total possible score is 5. If all 10 sections are completed the score is calculated and interpreted in percentage measures
Numeric Pain Rating Scale | follow up at 12th week
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes.

CONTACTS AND LOCATIONS:
Overall Officials: uneeb ur Rehman, MS*, Principal Investigator — Riphah International University
Locations (1):
- Al-Barkat Hospital, Gojra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balague F, Nordin M, Sheikhzadeh A, Echegoyen AC, Brisby H, Hoogewoud HM, Fredman P, Skovron ML. Recovery of severe sciatica. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2516-24. doi: 10.1097/00007632-199912010-00014. PMID 10626315
- [Background] Beurskens AJ, de Vet HC, Koke AJ, Lindeman E, Regtop W, van der Heijden GJ, Knipschild PG. Efficacy of traction for non-specific low back pain: a randomised clinical trial. Lancet. 1995 Dec 16;346(8990):1596-600. doi: 10.1016/s0140-6736(95)91930-9. PMID 7500752
- [Background] Bilgilisoy Filiz M, Kilic Z, Uckun A, Cakir T, Koldas Dogan S, Toraman NF. Mechanical Traction for Lumbar Radicular Pain: Supine or Prone? A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Jun;97(6):433-439. doi: 10.1097/PHM.0000000000000892. PMID 29309314
- [Background] Cai C, Pua YH, Lim KC. A clinical prediction rule for classifying patients with low back pain who demonstrate short-term improvement with mechanical lumbar traction. Eur Spine J. 2009 Apr;18(4):554-61. doi: 10.1007/s00586-009-0909-9. Epub 2009 Mar 3. PMID 19255792
- [Background] Carey TS, Freburger JK, Holmes GM, Castel L, Darter J, Agans R, Kalsbeek W, Jackman A. A long way to go: practice patterns and evidence in chronic low back pain care. Spine (Phila Pa 1976). 2009 Apr 1;34(7):718-24. doi: 10.1097/BRS.0b013e31819792b0. PMID 19282797
- [Background] Koldas Dogan S, Sonel Tur B, Kurtais Y, Atay MB. Comparison of three different approaches in the treatment of chronic low back pain. Clin Rheumatol. 2008 Jul;27(7):873-81. doi: 10.1007/s10067-007-0815-7. Epub 2008 Jan 11. PMID 18188660
- [Background] Fritz JM, Thackeray A, Childs JD, Brennan GP. A randomized clinical trial of the effectiveness of mechanical traction for sub-groups of patients with low back pain: study methods and rationale. BMC Musculoskelet Disord. 2010 Apr 30;11:81. doi: 10.1186/1471-2474-11-81. PMID 20433733
- [Background] Hahne AJ, Ford JJ, McMeeken JM. Conservative management of lumbar disc herniation with associated radiculopathy: a systematic review. Spine (Phila Pa 1976). 2010 May 15;35(11):E488-504. doi: 10.1097/BRS.0b013e3181cc3f56. PMID 20421859
- [Background] Hansen FR, Bendix T, Skov P, Jensen CV, Kristensen JH, Krohn L, Schioeler H. Intensive, dynamic back-muscle exercises, conventional physiotherapy, or placebo-control treatment of low-back pain. A randomized, observer-blind trial. Spine (Phila Pa 1976). 1993 Jan;18(1):98-108. doi: 10.1097/00007632-199301000-00015. PMID 8434332